CLINICAL TRIAL: NCT03333837
Title: IMOVE: Improvisational Movement for People With Memory Loss and Their Caregivers
Brief Title: Improvisational Movement for People With Memory Loss and Their Caregivers
Acronym: IMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00042460; R01AT009444 (NIH)
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer's Disease (Incl Subtypes); Dementia; Mild Cognitive Impairment
Keywords: Improvisation; Memory loss; Caregivers; Quality of Life; Dance; Social Group; MRI; mild cognitive impairment; MCI; Social engagement
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Memory Disorders | interventions — Social Group

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Investigators will use a 2x2 factorial design to test the separate and combined effects of social engagement and dance movement on QoL in 120 community-dwelling older adults adjudicated as having mild cognitive impairment (MCI) or early-stage dementia of the presumed AD or mixed AD/vascular type. Participants will be randomized to one of four 12-week interventions: 1) Dance Group 2) Non-group Dance, 3) Social Group, or 4) No Contact Control.
Who Masked: Outcomes Assessor
Masking Description: All study assessments will be conducted by experienced staff certified annually on the proper conduct of study assessments and blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dance Group (Active Comparator): The Dance Group will participate in 1-hour group improvisational dance lessons 2x/week for 12 weeks. Improvisational dance classes are grounded in 4 principles that shape the tone of the class and result in a sense of social belonging: non-judgment, non-competitiveness, curiosity, and playfulness. The following training strategies are used to maintain: active imagination, variability, and pacing.
  Interventions: Behavioral: Dance Group
- Non-group Dance (Active Comparator): The Non-group dance intervention is designed to capture the same dance movement and auditory stimuli as the group class without social interaction. Recordings of the dance instructor teaching a dance class will be played. This will ensure participants hear comparable music and receive comparable verbal auditory cues to prompt dance movements that students in the group class will hear, without interacting with other people. Improvisational dance is particularly suited for this means of delivery because the primary method of instruction is verbal auditory cueing. Participants will be asked to follow the same schedule as participants in the Dance Group arm and complete 2 one-hour dance sessions each week.
  Interventions: Behavioral: Non-Group Dance
- Social Group (Active Comparator): The social group will consist of improvisational party games to foster curiosity and playfulness, use imagery, and encourage non-judgment. Games that may be used include 'Balderdash', 'Wise and Otherwise', 'Charades', 'Pictionary', and 'Tell Me A Story' cards. These games will also use the same core strategies as the dance group. Games will be varied within an hour-long session to incorporate pacing and variability into the social group, akin to the dance group. The social group will occur 2x/week for 1 hour each time and be led by the same instructors who lead the Dance Group, to control for effects of personality of the group leader.
  Interventions: Behavioral: Social Group
- No Contact (Sham Comparator): A No Contact condition captures the condition of no added social contact and no added dance movement. Participants randomized to the No Contact condition will be asked to continue their current disease management and lifestyle for 12 weeks
  Interventions: Behavioral: No Contact

INTERVENTIONS:
Behavioral: Dance Group — Active imagination refers to working with imagery and is crucial in improvisatory practice. Verbal auditory cues are used to create movement scenarios that cue or activate the motor imagination. Variability means the improvisational method does not aim to learn a specific movement pattern and habituate to it. Cues are delivered quickly, one after another. Within an average of two minutes, tasks requiring quicker decision-making are introduced. Pacing is the rate at which new movement prompts are presented. Quick changes in pace avoid defaulting to habitual responses, thereby facilitating new movement options. Participants cannot rely on copying another, memory, or anticipation to address the motor problem.
  Arms: Dance Group
Behavioral: Non-Group Dance — The caregiver will be asked to stay in the area while the subject is dancing. A video camera will be affixed in an upper corner of the room to record individual dance sessions. This recording will yield data that a trained student or staff member can view and code to document movement fidelity (e.g., that the person has responded to the dance prompts and for the purpose of comparing the amount of quality of movements that occur in individual vs. group dance settings). For the first two sessions, study staff would observe the full dance session from outside the room to be sure that instruction was clear and adherence was attained, and that no safety issues arise.
  Arms: Non-group Dance
Behavioral: Social Group — The social group will consist of improvisational party games to foster curiosity and playfulness, use imagery, and encourage non-judgment. Games that may be used include 'Balderdash', 'Wise and Otherwise', 'Charades', 'Pictionary', and 'Tell Me A Story' cards. These games will also use the same core strategies as the dance group. Games will be varied within an hour-long session to incorporate pacing and variability into the social group, akin to the dance group. The social group will occur 2x/week for 1 hour each time and be led by the same instructors who lead the Dance Group, to control for effects of personality of the group leader.
  Arms: Social Group
Behavioral: No Contact — The condition of not receiving an intervention can have ethical implications and reduce retention rates. Therefore, these participants will be invited to join in a weekly community improvisational dance class after they complete the study, for as many sessions as they would like.
  Arms: No Contact

SUMMARY:
Dementia is a progressive decline in cognition that impairs a person's ability to perform activities of daily living. Changes in mood, gait, and balance are prominent secondary symptoms of Alzheimer's dementia that can dramatically decrease quality of life for the person with dementia and increase caregiver burden. The overall aim of this study is to determine the independent and combined effects of dance movement and social engagement on quality of life in people with early-stage dementia, and test the neural mechanisms of these effects.

DETAILED DESCRIPTION:
Dementia is a progressive decline in cognition that impairs a person's ability to perform activities of daily living. Alzheimer's disease is the most common form of dementia, the most common neurodegenerative disease in older adults, and the 6th leading cause of death in the US. Neuropsychiatric symptoms (apathy, depression, anxiety) and altered gait and balance are prominent secondary symptoms of Alzheimer's disease that increase medical costs and decrease quality of life for both the person with dementia and their caregiver.

In a report from the Secretariat (Executive Board, 134th Session, December 20th, 2013), the World Health Organization identified a need to integrate evidence-based palliative care services into the continuum of care for serious chronic diseases, including Alzheimer's disease. However, two recent NIH workshops identified major gaps in the evidence supporting the wider use of non-pharmacologic activities to ameliorate secondary symptoms of chronic disease. Arts-based activities were identified as particularly understudied for symptom management, given growing evidence that various arts-based activities can improve quality of life, relieve symptoms, and reduce reliance on medications. It is important that these benefits can be achieved without adding medications. Dance is an arts-based activity that can improve quality of life, decrease symptoms of depression, and improve balance in healthy older adults, those with Parkinson disease, and Alzheimer's disease. Thus, dance is a non-pharmacological intervention that simultaneously addresses two sets of prominent secondary symptoms in Alzheimer's disease: 1) gait and balance and 2) neuropsychiatric symptoms. However, the mechanisms through which dance exerts these effects are unknown.

Pilot data from the investigators' laboratory suggest that participating in a group improvisational movement class twice weekly improved balance and connectivity in motor-related brain regions, as well as improving mood and connectivity in brain regions associated with social engagement. Improvisation is the ability to create new gestures and movements spontaneously. Improvisation can be a part of many different art forms. However, improvisational movement can also be practiced as a specific dance form. The objective in improvisational movement is that choreographed movement is replaced by a cue or prompt that allows the possibility for multiple responses. This unique form of dance is especially well-suited for people with dementia because it: 1) does not rely heavily on memory of repeated movements; 2) can be seamlessly adapted to include sitting, standing, or moving around the room; 3) is cognitively challenging; and 4) fosters a social, playful atmosphere. Participants seemed to benefit from both the social nature of the class and the movement. Therefore, the overall aim of this proposal is to experimentally determine the independent and combined effects of dance movement and social engagement on quality of life in people with early stage dementia, and test the neural mechanisms of these effects.

To accomplish this goal, the investigators will use a 2x2 factorial design and randomize 120 community-dwelling older adults adjudicated as having early-stage dementia of the presumed Alzheimer's type to one of four 3-month interventions: 1) Dance Group, 2) Non-group Dance, 3) Social Group, or 4) No Contact Control.

It is not hypothesized that dance affects the underlying disease course, and therefore no improvement is expected in cognition.

ELIGIBILITY:
Inclusion Criteria:

Age 60-85 years

Adjudicated as having mild cognitive impairment or early-stage dementia of Alzheimer's, vascular, or mixed Alzheimer's/vascular type

MRI compatible

English speaking

Have study partner who is around the person with dementia approximately 10 hours/week and is willing to be an active study partner.

Able to attend bi-weekly intervention classes or come to study visits for no-contact control.

Not enrolled in another interventional study for at least 3 months prior to beginning this study.

Exclusion Criteria:

Untreated depression

Other causes of dementia (for example, frontotemporal, early onset, Lewy body or Parkinsonian dementia)

Current cancer treatment or other major medical problems that might independently affect cognition or movement

Other neurological disorders (e.g., Parkinson disease, multiple sclerosis)

Taking medication that could negatively influence safety during intervention

Planned extensive travel during the study period

Any reason for which the study doctor or personal physician feels the intervention is contraindicated for the participant

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hugenschmidt, PhD, Principal Investigator — Assistant Professor Gerontology and Geriatric Medicine
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer's Association. 2013 Alzheimer's disease facts and figures. Alzheimers Dement. 2013 Mar;9(2):208-45. doi: 10.1016/j.jalz.2013.02.003. PMID 23507120
- [Background] Gaugler JE, Yu F, Krichbaum K, Wyman JF. Predictors of nursing home admission for persons with dementia. Med Care. 2009 Feb;47(2):191-8. doi: 10.1097/MLR.0b013e31818457ce. PMID 19169120
- [Background] Okura T, Langa KM. Caregiver burden and neuropsychiatric symptoms in older adults with cognitive impairment: the Aging, Demographics, and Memory Study (ADAMS). Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):116-21. doi: 10.1097/WAD.0b013e318203f208. PMID 21192239
- [Background] Schubert CC, Boustani M, Callahan CM, Perkins AJ, Hui S, Hendrie HC. Acute care utilization by dementia caregivers within urban primary care practices. J Gen Intern Med. 2008 Nov;23(11):1736-40. doi: 10.1007/s11606-008-0711-0. Epub 2008 Aug 9. PMID 18690489
- [Background] Committee, S.o.t.F., State of the Field Report: Arts in Healthcare 2009, 2009, Society for the Arts in Healthcare: Washington, DC.
- [Background] Verghese J, Lipton RB, Katz MJ, Hall CB, Derby CA, Kuslansky G, Ambrose AF, Sliwinski M, Buschke H. Leisure activities and the risk of dementia in the elderly. N Engl J Med. 2003 Jun 19;348(25):2508-16. doi: 10.1056/NEJMoa022252. PMID 12815136
- [Background] Verghese J. Cognitive and mobility profile of older social dancers. J Am Geriatr Soc. 2006 Aug;54(8):1241-4. doi: 10.1111/j.1532-5415.2006.00808.x. PMID 16913992
- [Background] Coubard OA, Duretz S, Lefebvre V, Lapalus P, Ferrufino L. Practice of contemporary dance improves cognitive flexibility in aging. Front Aging Neurosci. 2011 Sep 20;3:13. doi: 10.3389/fnagi.2011.00013. eCollection 2011. PMID 21960971
- [Background] Earhart GM. Dance as therapy for individuals with Parkinson disease. Eur J Phys Rehabil Med. 2009 Jun;45(2):231-8. PMID 19532110
- [Background] Hackney, M.E., S. Kantorovich, and G.M. Earhart, A study of the effects of Argentine tango as a form of partnered dance for those with Parkinson disease and the healthy elderly. American Journal of Dance Therapy, 2007. 29(2): p. 109-127.
- [Background] Hui E, Chui BT, Woo J. Effects of dance on physical and psychological well-being in older persons. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):e45-50. doi: 10.1016/j.archger.2008.08.006. Epub 2008 Oct 5. PMID 18838181
- [Background] Shanahan J, Morris ME, Bhriain ON, Saunders J, Clifford AM. Dance for people with Parkinson disease: what is the evidence telling us? Arch Phys Med Rehabil. 2015 Jan;96(1):141-53. doi: 10.1016/j.apmr.2014.08.017. Epub 2014 Sep 16. PMID 25223491
- [Background] Sharp K, Hewitt J. Dance as an intervention for people with Parkinson's disease: a systematic review and meta-analysis. Neurosci Biobehav Rev. 2014 Nov;47:445-56. doi: 10.1016/j.neubiorev.2014.09.009. Epub 2014 Sep 28. PMID 25268548
- [Background] Tjaden K. Speech and Swallowing in Parkinson's Disease. Top Geriatr Rehabil. 2008;24(2):115-126. doi: 10.1097/01.TGR.0000318899.87690.44. PMID 19946386
- [Background] Adam D, Ramli A, Shahar S. Effectiveness of a Combined Dance and Relaxation Intervention on Reducing Anxiety and Depression and Improving Quality of Life among the Cognitively Impaired Elderly. Sultan Qaboos Univ Med J. 2016 Feb;16(1):e47-53. doi: 10.18295/squmj.2016.16.01.009. Epub 2016 Feb 2. PMID 26909213
- [Background] Guzman-Garcia A, Mukaetova-Ladinska E, James I. Introducing a Latin ballroom dance class to people with dementia living in care homes, benefits and concerns: a pilot study. Dementia (London). 2013 Sep;12(5):523-35. doi: 10.1177/1471301211429753. Epub 2012 Mar 16. PMID 24337327
- [Background] Roepke SK, Allison M, Von Kanel R, Mausbach BT, Chattillion EA, Harmell AL, Patterson TL, Dimsdale JE, Mills PJ, Ziegler MG, Ancoli-Israel S, Grant I. Relationship between chronic stress and carotid intima-media thickness (IMT) in elderly Alzheimer's disease caregivers. Stress. 2012 Mar;15(2):121-9. doi: 10.3109/10253890.2011.596866. Epub 2011 Jul 26. PMID 21790484
- [Background] Gouin JP, Glaser R, Malarkey WB, Beversdorf D, Kiecolt-Glaser J. Chronic stress, daily stressors, and circulating inflammatory markers. Health Psychol. 2012 Mar;31(2):264-8. doi: 10.1037/a0025536. Epub 2011 Sep 19. PMID 21928900
- [Background] von Kanel R, Mausbach BT, Dimsdale JE, Mills PJ, Patterson TL, Ancoli-Israel S, Ziegler MG, Roepke SK, Chattillion EA, Allison M, Grant I. Effect of chronic dementia caregiving and major transitions in the caregiving situation on kidney function: a longitudinal study. Psychosom Med. 2012 Feb-Mar;74(2):214-20. doi: 10.1097/PSY.0b013e3182408c14. Epub 2012 Jan 27. PMID 22286846
- [Background] von Kanel R, Mills PJ, Mausbach BT, Dimsdale JE, Patterson TL, Ziegler MG, Ancoli-Israel S, Allison M, Chattillion EA, Grant I. Effect of Alzheimer caregiving on circulating levels of C-reactive protein and other biomarkers relevant to cardiovascular disease risk: a longitudinal study. Gerontology. 2012;58(4):354-65. doi: 10.1159/000334219. Epub 2011 Nov 29. PMID 22133914
- [Background] Mausbach BT, Chattillion E, Roepke SK, Ziegler MG, Milic M, von Kanel R, Dimsdale JE, Mills PJ, Patterson TL, Allison MA, Ancoli-Israel S, Grant I. A longitudinal analysis of the relations among stress, depressive symptoms, leisure satisfaction, and endothelial function in caregivers. Health Psychol. 2012 Jul;31(4):433-40. doi: 10.1037/a0027783. Epub 2012 Apr 9. PMID 22486550
- [Background] Chattillion EA, Mausbach BT, Roepke SK, von Kanel R, Mills PJ, Dimsdale JE, Allison M, Ziegler MG, Patterson TL, Ancoli-Israel S, Grant I. Leisure activities, caregiving demands and catecholamine levels in dementia caregivers. Psychol Health. 2012;27(10):1134-49. doi: 10.1080/08870446.2011.637559. Epub 2011 Dec 12. PMID 22149759
- [Background] Christakis NA, Allison PD. Mortality after the hospitalization of a spouse. N Engl J Med. 2006 Feb 16;354(7):719-30. doi: 10.1056/NEJMsa050196. PMID 16481639
- [Background] Harvey L, Mitchell R, Brodaty H, Draper B, Close J. The influence of dementia on injury-related hospitalisations and outcomes in older adults. Injury. 2016 Jan;47(1):226-34. doi: 10.1016/j.injury.2015.09.021. Epub 2015 Oct 9. PMID 26534784
- [Background] van Doorn C, Gruber-Baldini AL, Zimmerman S, Hebel JR, Port CL, Baumgarten M, Quinn CC, Taler G, May C, Magaziner J; Epidemiology of Dementia in Nursing Homes Research Group. Dementia as a risk factor for falls and fall injuries among nursing home residents. J Am Geriatr Soc. 2003 Sep;51(9):1213-8. doi: 10.1046/j.1532-5415.2003.51404.x. PMID 12919232
- [Background] Tchalla AE, Dufour AB, Travison TG, Habtemariam D, Iloputaife I, Manor B, Lipsitz LA. Patterns, predictors, and outcomes of falls trajectories in older adults: the MOBILIZE Boston Study with 5 years of follow-up. PLoS One. 2014 Sep 3;9(9):e106363. doi: 10.1371/journal.pone.0106363. eCollection 2014. PMID 25184785
- [Background] Taylor ME, Delbaere K, Lord SR, Mikolaizak AS, Brodaty H, Close JC. Neuropsychological, physical, and functional mobility measures associated with falls in cognitively impaired older adults. J Gerontol A Biol Sci Med Sci. 2014 Aug;69(8):987-95. doi: 10.1093/gerona/glt166. Epub 2013 Oct 22. PMID 24149433
- [Background] McGough EL, Logsdon RG, Kelly VE, Teri L. Functional mobility limitations and falls in assisted living residents with dementia: physical performance assessment and quantitative gait analysis. J Geriatr Phys Ther. 2013 Apr-Jun;36(2):78-86. doi: 10.1519/JPT.0b013e318268de7f. PMID 22976811
- [Background] Bruce-Keller AJ, Brouillette RM, Tudor-Locke C, Foil HC, Gahan WP, Nye DM, Guillory L, Keller JN. Relationship between cognitive domains, physical performance, and gait in elderly and demented subjects. J Alzheimers Dis. 2012;30(4):899-908. doi: 10.3233/JAD-2012-120025. PMID 22466001
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Szczepanska-Gieracha J, Cieslik B, Chamela-Bilinska D, Kuczynski M. Postural Stability of Elderly People With Cognitive Impairments. Am J Alzheimers Dis Other Demen. 2016 May;31(3):241-6. doi: 10.1177/1533317515602547. Epub 2015 Sep 17. PMID 26385944
- [Background] Cedervall Y, Halvorsen K, Aberg AC. A longitudinal study of gait function and characteristics of gait disturbance in individuals with Alzheimer's disease. Gait Posture. 2014 Apr;39(4):1022-7. doi: 10.1016/j.gaitpost.2013.12.026. Epub 2014 Jan 21. PMID 24491520
- [Background] Dodge HH, Mattek NC, Austin D, Hayes TL, Kaye JA. In-home walking speeds and variability trajectories associated with mild cognitive impairment. Neurology. 2012 Jun 12;78(24):1946-52. doi: 10.1212/WNL.0b013e318259e1de. PMID 22689734
- [Background] Buracchio T, Dodge HH, Howieson D, Wasserman D, Kaye J. The trajectory of gait speed preceding mild cognitive impairment. Arch Neurol. 2010 Aug;67(8):980-6. doi: 10.1001/archneurol.2010.159. PMID 20697049
- [Background] Fitzpatrick AL, Buchanan CK, Nahin RL, Dekosky ST, Atkinson HH, Carlson MC, Williamson JD; Ginkgo Evaluation of Memory (GEM) Study Investigators. Associations of gait speed and other measures of physical function with cognition in a healthy cohort of elderly persons. J Gerontol A Biol Sci Med Sci. 2007 Nov;62(11):1244-51. doi: 10.1093/gerona/62.11.1244. PMID 18000144
- [Background] Kuo HK, Leveille SG, Yu YH, Milberg WP. Cognitive function, habitual gait speed, and late-life disability in the National Health and Nutrition Examination Survey (NHANES) 1999-2002. Gerontology. 2007;53(2):102-10. doi: 10.1159/000096792. Epub 2006 Nov 6. PMID 17090975
- [Background] Nadkarni NK, Nunley KA, Aizenstein H, Harris TB, Yaffe K, Satterfield S, Newman AB, Rosano C; Health ABC Study. Association between cerebellar gray matter volumes, gait speed, and information-processing ability in older adults enrolled in the Health ABC study. J Gerontol A Biol Sci Med Sci. 2014 Aug;69(8):996-1003. doi: 10.1093/gerona/glt151. Epub 2013 Oct 29. PMID 24170673
- [Background] Verghese J, Annweiler C, Ayers E, Barzilai N, Beauchet O, Bennett DA, Bridenbaugh SA, Buchman AS, Callisaya ML, Camicioli R, Capistrant B, Chatterji S, De Cock AM, Ferrucci L, Giladi N, Guralnik JM, Hausdorff JM, Holtzer R, Kim KW, Kowal P, Kressig RW, Lim JY, Lord S, Meguro K, Montero-Odasso M, Muir-Hunter SW, Noone ML, Rochester L, Srikanth V, Wang C. Motoric cognitive risk syndrome: multicountry prevalence and dementia risk. Neurology. 2014 Aug 19;83(8):718-26. doi: 10.1212/WNL.0000000000000717. Epub 2014 Jul 16. PMID 25031288
- [Background] Verghese J, Wang C, Lipton RB, Holtzer R. Motoric cognitive risk syndrome and the risk of dementia. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):412-8. doi: 10.1093/gerona/gls191. Epub 2012 Sep 17. PMID 22987797
- [Background] Watson NL, Rosano C, Boudreau RM, Simonsick EM, Ferrucci L, Sutton-Tyrrell K, Hardy SE, Atkinson HH, Yaffe K, Satterfield S, Harris TB, Newman AB; Health ABC Study. Executive function, memory, and gait speed decline in well-functioning older adults. J Gerontol A Biol Sci Med Sci. 2010 Oct;65(10):1093-100. doi: 10.1093/gerona/glq111. Epub 2010 Jun 25. PMID 20581339
- [Background] Gietzelt M, Wolf KH, Kohlmann M, Marschollek M, Haux R. Measurement of accelerometry-based gait parameters in people with and without dementia in the field: a technical feasibility study. Methods Inf Med. 2013;52(4):319-25. doi: 10.3414/ME12-02-0009. Epub 2013 Jun 28. PMID 23807731
- [Background] Verghese J, Wang C, Lipton RB, Holtzer R, Xue X. Quantitative gait dysfunction and risk of cognitive decline and dementia. J Neurol Neurosurg Psychiatry. 2007 Sep;78(9):929-35. doi: 10.1136/jnnp.2006.106914. Epub 2007 Jan 19. PMID 17237140
- [Background] Ohman H, Savikko N, Strandberg T, Kautiainen H, Raivio M, Laakkonen ML, Tilvis R, Pitkala KH. Effects of Exercise on Functional Performance and Fall Rate in Subjects with Mild or Advanced Alzheimer's Disease: Secondary Analyses of a Randomized Controlled Study. Dement Geriatr Cogn Disord. 2016;41(3-4):233-41. doi: 10.1159/000445712. Epub 2016 May 10. PMID 27160164
- [Background] Del Campo N, Payoux P, Djilali A, Delrieu J, Hoogendijk EO, Rolland Y, Cesari M, Weiner MW, Andrieu S, Vellas B; MAPT/DSA Study Group. Relationship of regional brain beta-amyloid to gait speed. Neurology. 2016 Jan 5;86(1):36-43. doi: 10.1212/WNL.0000000000002235. Epub 2015 Dec 7. PMID 26643548
- [Background] Olazaran J, Hernandez-Tamames JA, Molina E, Garcia-Polo P, Dobato JL, Alvarez-Linera J, Martinez-Martin P; AD Research Unit Investigators. Clinical and anatomical correlates of gait dysfunction in Alzheimer's disease. J Alzheimers Dis. 2013;33(2):495-505. doi: 10.3233/JAD-2012-121207. PMID 23011219
- [Background] Regan B, Varanelli L. Adjustment, depression, and anxiety in mild cognitive impairment and early dementia: a systematic review of psychological intervention studies. Int Psychogeriatr. 2013 Dec;25(12):1963-84. doi: 10.1017/S104161021300152X. Epub 2013 Oct 14. PMID 24125507
- [Background] Zhang JG, Ishikawa-Takata K, Yamazaki H, Morita T, Ohta T. Postural stability and physical performance in social dancers. Gait Posture. 2008 May;27(4):697-701. doi: 10.1016/j.gaitpost.2007.09.004. Epub 2007 Nov 5. PMID 17981468
- [Background] Hackney ME, Byers C, Butler G, Sweeney M, Rossbach L, Bozzorg A. Adapted Tango Improves Mobility, Motor-Cognitive Function, and Gait but Not Cognition in Older Adults in Independent Living. J Am Geriatr Soc. 2015 Oct;63(10):2105-13. doi: 10.1111/jgs.13650. Epub 2015 Oct 12. PMID 26456371
- [Background] Fernandez-Arguelles EL, Rodriguez-Mansilla J, Antunez LE, Garrido-Ardila EM, Munoz RP. Effects of dancing on the risk of falling related factors of healthy older adults: a systematic review. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):1-8. doi: 10.1016/j.archger.2014.10.003. Epub 2014 Nov 6. PMID 25456888
- [Background] Eyigor S, Karapolat H, Durmaz B, Ibisoglu U, Cakir S. A randomized controlled trial of Turkish folklore dance on the physical performance, balance, depression and quality of life in older women. Arch Gerontol Geriatr. 2009 Jan-Feb;48(1):84-8. doi: 10.1016/j.archger.2007.10.008. Epub 2008 Feb 20. PMID 18068829
- [Background] Haboush, A., et al., Ballroom dance lessons for geriatric depression: An exploratory study. The Arts in Psychotherapy, 2006. 33(2): p. 89-97.
- [Background] Mavrovouniotis FH, Argiriadou EA, Papaioannou CS. Greek traditional dances and quality of old people's life. J Bodyw Mov Ther. 2010 Jul;14(3):209-18. doi: 10.1016/j.jbmt.2008.11.005. Epub 2009 Feb 7. PMID 20538217
- [Background] Brauninger, I., The efficacy of dance movement therapy group on improvement of quality of life: A randomized controlled trial. The Arts in Psychotherapy, 2012. 39: p. 296-303.
- [Background] Abreu M, Hartley G. The effects of Salsa dance on balance, gait, and fall risk in a sedentary patient with Alzheimer's dementia, multiple comorbidities, and recurrent falls. J Geriatr Phys Ther. 2013 Apr-Jun;36(2):100-8. doi: 10.1519/JPT.0b013e318267aa54. PMID 22955042
- [Background] Goldman, D., I want to be ready: Improvised dance as a practice of freedom. 2010, Ann Arbor, MI: University of Michigan Press.
- [Background] Montuori, A., The complexity of improvisation and the improvisation of complexity: Social science, art and creativity. Human Relations, 2003. 56(2): p. 237-255.
- [Background] Lockford, L. and R. Pelias, Bodily poeticizing in theatrical improvisation: A typology of performative knowledge. Theatre Topics, 2004. 14(2): p. 431-443.
- [Background] Sawyer, R., Improvisation and the creative process: Dewey, Collingwood, and the aesthetics of spontaneity. Journal of Aesthetics and Art Criticism, 2000. 58(2): p. 149-161.
- [Background] Batson, G., et al., Effects of improvisational dance on balance in Parkinson's disease: A two-phase fMRI case study. Physical and Occupational Therapy in Geriatrics, 2014. 32(3): p. 188-197.
- [Background] Batson G, Hugenschmidt CE, Soriano CT. Verbal Auditory Cueing of Improvisational Dance: A Proposed Method for Training Agency in Parkinson's Disease. Front Neurol. 2016 Feb 17;7:15. doi: 10.3389/fneur.2016.00015. eCollection 2016. PMID 26925029
- [Background] Weintraub S, Salmon D, Mercaldo N, Ferris S, Graff-Radford NR, Chui H, Cummings J, DeCarli C, Foster NL, Galasko D, Peskind E, Dietrich W, Beekly DL, Kukull WA, Morris JC. The Alzheimer's Disease Centers' Uniform Data Set (UDS): the neuropsychologic test battery. Alzheimer Dis Assoc Disord. 2009 Apr-Jun;23(2):91-101. doi: 10.1097/WAD.0b013e318191c7dd. PMID 19474567
- [Background] Alberici A, Benussi A, Premi E, Borroni B, Padovani A. Clinical, genetic, and neuroimaging features of Early Onset Alzheimer Disease: the challenges of diagnosis and treatment. Curr Alzheimer Res. 2014;11(10):909-17. doi: 10.2174/1567205011666141107151606. PMID 25387334
- [Background] Dziak, J.J., L.M. Collins, and A.T. Wagner, FactorialPowerPlan SAS macro suite users' guide (Version 1.0). University Park: The Methodology Center, Penn State, 2013. Retrieved from http://methodology.psy.edu.
- [Background] Petzinger GM, Fisher BE, McEwen S, Beeler JA, Walsh JP, Jakowec MW. Exercise-enhanced neuroplasticity targeting motor and cognitive circuitry in Parkinson's disease. Lancet Neurol. 2013 Jul;12(7):716-26. doi: 10.1016/S1474-4422(13)70123-6. PMID 23769598
- [Background] Duncan RP, Earhart GM. Randomized controlled trial of community-based dancing to modify disease progression in Parkinson disease. Neurorehabil Neural Repair. 2012 Feb;26(2):132-43. doi: 10.1177/1545968311421614. Epub 2011 Sep 29. PMID 21959675
- [Background] Barrios H, Narciso S, Guerreiro M, Maroco J, Logsdon R, de Mendonca A. Quality of life in patients with mild cognitive impairment. Aging Ment Health. 2013;17(3):287-92. doi: 10.1080/13607863.2012.747083. Epub 2012 Dec 7. PMID 23215827
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Logsdon RG, McCurry SM, Teri L. Evidence-Based Interventions to Improve Quality of Life for Individuals with Dementia. Alzheimers care today. 2007;8(4):309-318. PMID 19030120
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] McHorney CA, Ware JE Jr, Rogers W, Raczek AE, Lu JF. The validity and relative precision of MOS short- and long-form health status scales and Dartmouth COOP charts. Results from the Medical Outcomes Study. Med Care. 1992 May;30(5 Suppl):MS253-65. doi: 10.1097/00005650-199205001-00025. PMID 1583937
- [Background] Rose DJ, Lucchese N, Wiersma LD. Development of a multidimensional balance scale for use with functionally independent older adults. Arch Phys Med Rehabil. 2006 Nov;87(11):1478-85. doi: 10.1016/j.apmr.2006.07.263. PMID 17084123
- [Background] Norris JA, Marsh AP, Smith IJ, Kohut RI, Miller ME. Ability of static and statistical mechanics posturographic measures to distinguish between age and fall risk. J Biomech. 2005 Jun;38(6):1263-72. doi: 10.1016/j.jbiomech.2004.06.014. PMID 15863111
- [Background] Brauer SG, Burns YR, Galley P. A prospective study of laboratory and clinical measures of postural stability to predict community-dwelling fallers. J Gerontol A Biol Sci Med Sci. 2000 Aug;55(8):M469-76. doi: 10.1093/gerona/55.8.m469. PMID 10952371
- [Background] Hahn ME, Chou LS. Can motion of individual body segments identify dynamic instability in the elderly? Clin Biomech (Bristol). 2003 Oct;18(8):737-44. doi: 10.1016/s0268-0033(03)00139-6. PMID 12957560
- [Background] Mak MK, Ng PL. Mediolateral sway in single-leg stance is the best discriminator of balance performance for Tai-Chi practitioners. Arch Phys Med Rehabil. 2003 May;84(5):683-6. doi: 10.1016/s0003-9993(02)04810-4. PMID 12736881
- [Background] Maki BE, Holliday PJ, Topper AK. A prospective study of postural balance and risk of falling in an ambulatory and independent elderly population. J Gerontol. 1994 Mar;49(2):M72-84. doi: 10.1093/geronj/49.2.m72. PMID 8126355
- [Background] Mitchell SL, Collins JJ, De Luca CJ, Burrows A, Lipsitz LA. Open-loop and closed-loop postural control mechanisms in Parkinson's disease: increased mediolateral activity during quiet standing. Neurosci Lett. 1995 Sep 8;197(2):133-6. doi: 10.1016/0304-3940(95)11924-l. PMID 8552278
- [Background] Laughton CA, Slavin M, Katdare K, Nolan L, Bean JF, Kerrigan DC, Phillips E, Lipsitz LA, Collins JJ. Aging, muscle activity, and balance control: physiologic changes associated with balance impairment. Gait Posture. 2003 Oct;18(2):101-8. doi: 10.1016/s0966-6362(02)00200-x. PMID 14654213
- [Background] Beauchet O, Freiberger E, Annweiler C, Kressig RW, Herrmann FR, Allali G. Test-retest reliability of stride time variability while dual tasking in healthy and demented adults with frontotemporal degeneration. J Neuroeng Rehabil. 2011 Jul 11;8(1):37. doi: 10.1186/1743-0003-8-37. PMID 21745370
- [Background] Dubost V, Kressig RW, Gonthier R, Herrmann FR, Aminian K, Najafi B, Beauchet O. Relationships between dual-task related changes in stride velocity and stride time variability in healthy older adults. Hum Mov Sci. 2006 Jun;25(3):372-82. doi: 10.1016/j.humov.2006.03.004. Epub 2006 May 22. PMID 16714067
- [Background] Mijnarends DM, Meijers JM, Halfens RJ, ter Borg S, Luiking YC, Verlaan S, Schoberer D, Cruz Jentoft AJ, van Loon LJ, Schols JM. Validity and reliability of tools to measure muscle mass, strength, and physical performance in community-dwelling older people: a systematic review. J Am Med Dir Assoc. 2013 Mar;14(3):170-8. doi: 10.1016/j.jamda.2012.10.009. Epub 2012 Dec 29. PMID 23276432
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] Simonsick EM, Newman AB, Nevitt MC, Kritchevsky SB, Ferrucci L, Guralnik JM, Harris T; Health ABC Study Group. Measuring higher level physical function in well-functioning older adults: expanding familiar approaches in the Health ABC study. J Gerontol A Biol Sci Med Sci. 2001 Oct;56(10):M644-9. doi: 10.1093/gerona/56.10.m644. PMID 11584038
- [Background] Houston DK, Leng X, Bray GA, Hergenroeder AL, Hill JO, Jakicic JM, Johnson KC, Neiberg RH, Marsh AP, Rejeski WJ, Kritchevsky SB; Action for Health In Diabetes (Look AHEAD) Movement and Memory Ancillary Study Research Group. A long-term intensive lifestyle intervention and physical function: the look AHEAD Movement and Memory Study. Obesity (Silver Spring). 2015 Jan;23(1):77-84. doi: 10.1002/oby.20944. Epub 2014 Nov 29. PMID 25452229
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Costa, P.T. and R.R. McCrae, The NEO-PI/NEO-FFI manual supplement. 1989, Odessa, FL: Psychological Assessment Resources.
- [Background] Orgeta V, Leung P. Personality and dementia caring: a review and commentary. Curr Opin Psychiatry. 2015 Jan;28(1):57-65. doi: 10.1097/YCO.0000000000000116. PMID 25420192
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Lueken U, Seidl U, Volker L, Schweiger E, Kruse A, Schroder J. Development of a short version of the Apathy Evaluation Scale specifically adapted for demented nursing home residents. Am J Geriatr Psychiatry. 2007 May;15(5):376-85. doi: 10.1097/JGP.0b013e3180437db3. PMID 17463188
- [Background] Cardaciotto L, Herbert JD, Forman EM, Moitra E, Farrow V. The assessment of present-moment awareness and acceptance: the Philadelphia Mindfulness Scale. Assessment. 2008 Jun;15(2):204-23. doi: 10.1177/1073191107311467. Epub 2008 Jan 9. PMID 18187399
- [Background] Kattenstroth JC, Kolankowska I, Kalisch T, Dinse HR. Superior sensory, motor, and cognitive performance in elderly individuals with multi-year dancing activities. Front Aging Neurosci. 2010 Jul 21;2:31. doi: 10.3389/fnagi.2010.00031. eCollection 2010. PMID 20725636
- [Background] Kattenstroth JC, Kalisch T, Holt S, Tegenthoff M, Dinse HR. Six months of dance intervention enhances postural, sensorimotor, and cognitive performance in elderly without affecting cardio-respiratory functions. Front Aging Neurosci. 2013 Feb 26;5:5. doi: 10.3389/fnagi.2013.00005. eCollection 2013. PMID 23447455
- [Background] Kattenstroth, J.C., et al., Dance Therapy for Cognitive Enhancement in the Elderly. Journal of Psychophysiology, 2011. 25: p. 17-17.
- [Background] Bollen, K.A., Structural equations with latent variables. 1989, Hoboken, NJ: Wiley.
- [Background] Bizik G, Picard M, Nijjar R, Tourjman V, McEwen BS, Lupien SJ, Juster RP. Allostatic load as a tool for monitoring physiological dysregulations and comorbidities in patients with severe mental illnesses. Harv Rev Psychiatry. 2013 Nov-Dec;21(6):296-313. doi: 10.1097/HRP.0000000000000012. PMID 24201821
- [Background] McEwen BS. Brain on stress: how the social environment gets under the skin. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17180-5. doi: 10.1073/pnas.1121254109. Epub 2012 Oct 8. PMID 23045648
- [Background] McEwen BS, Stellar E. Stress and the individual. Mechanisms leading to disease. Arch Intern Med. 1993 Sep 27;153(18):2093-101. PMID 8379800
- [Background] Wahbeh H, Kishiyama SS, Zajdel D, Oken BS. Salivary cortisol awakening response in mild Alzheimer disease, caregivers, and noncaregivers. Alzheimer Dis Assoc Disord. 2008 Apr-Jun;22(2):181-3. doi: 10.1097/WAD.0b013e31815a9dff. PMID 18525292
- [Background] de Vugt ME, Nicolson NA, Aalten P, Lousberg R, Jolle J, Verhey FR. Behavioral problems in dementia patients and salivary cortisol patterns in caregivers. J Neuropsychiatry Clin Neurosci. 2005 Spring;17(2):201-7. doi: 10.1176/jnp.17.2.201. PMID 15939974
- [Background] Danucalov MA, Kozasa EH, Ribas KT, Galduroz JC, Garcia MC, Verreschi IT, Oliveira KC, Romani de Oliveira L, Leite JR. A yoga and compassion meditation program reduces stress in familial caregivers of Alzheimer's disease patients. Evid Based Complement Alternat Med. 2013;2013:513149. doi: 10.1155/2013/513149. Epub 2013 Apr 18. PMID 23690846
- [Background] Ornish D, Lin J, Chan JM, Epel E, Kemp C, Weidner G, Marlin R, Frenda SJ, Magbanua MJM, Daubenmier J, Estay I, Hills NK, Chainani-Wu N, Carroll PR, Blackburn EH. Effect of comprehensive lifestyle changes on telomerase activity and telomere length in men with biopsy-proven low-risk prostate cancer: 5-year follow-up of a descriptive pilot study. Lancet Oncol. 2013 Oct;14(11):1112-1120. doi: 10.1016/S1470-2045(13)70366-8. Epub 2013 Sep 17. PMID 24051140
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Derived] Thumuluri D, Lyday R, Babcock P, Ip EH, Kraft RA, Laurienti PJ, Barnstaple R, Soriano CT, Hugenschmidt CE. Improvisational Movement to Improve Quality of Life in Older Adults With Early-Stage Dementia: A Pilot Study. Front Sports Act Living. 2022 Jan 14;3:796101. doi: 10.3389/fspor.2021.796101. eCollection 2021. PMID 35098120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Persons With Dementia (PWDs) were enrolled with one caregiver each. There was never a time when one was enrolled without the other, so these two people are represented in the participant flow as a dyad.
Pre-assignment Details: Participants were enrolled in dyads consisting of one person with dementia (PWD) and one caregiver (CG). Participant flow section includes numbers as dyad since both were considered enrolled. Elsewhere in the record, numbers include either participants with dementia or caregivers as indicated in baseline analysis population description and in outcome titles or descriptions.
Groups:
- Never Randomized: Subject dyads who signed consent but withdrew prior to randomization.
Period: Overall Study
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact | Never Randomized
Started (Shows number of dyads who signed consent. Total number of participants is double the number of dyads. e.g., 20 dyads noted here = 40 participants) | 24 | 25 | 27 | 25 | 3
Completed (Shows number of dyads. Total number of participants is double the number of dyads. e.g., 20 dyads noted here = 40 participants) | 22 | 22 | 22 | 23 | 0
Not Completed | 2 | 3 | 5 | 2 | 3
Not completed — Adverse Event | 2 | 1 | 1 | 1 | 0
Not completed — Caregiver withdrew | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 3
Not completed — COVID interrupted enrollment--had to rescreen and didn't qualify | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis population included only the PWD portion of the dyad. No data for baseline analysis for caregivers was collected so it is not represented in this section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact | Never Randomized | Total
Number analyzed (Participants) | 24 | 25 | 27 | 25 | 3 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.33 (5.94) | 73.62 (7.10) | 76.75 (6.29) | 76.0 (6.43) | 69.87 (3.23) | 75.29 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 14 | 11 | 0 | 50
  Male | 12 | 12 | 13 | 14 | 3 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 27 | 25 | 3 | 103
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 6 | 2 | 0 | 13
  White | 21 | 22 | 20 | 23 | 3 | 89
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 27 | 25 | 3 | 104

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life in Alzheimer's Disease (QOL-AD)--Participants With Dementia (PWD)
Description: Self-reported quality of life in the person with dementia is the primary outcome and will be measured using the QOL-AD . The QOL-AD is validated for use in people with Mini Mental State Exam scores as low as 10.The QOL_AD contains 13 items.Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.The total score is the sum of all 13 item (range 13- 52) higher scores represent better outcomes.
Time Frame: Baseline
Population: Results at baseline for this outcome represent all PWD who were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 35.42 (5.02) | 38.10 (4.60) | 35.56 (4.15) | 36.12 (5.75)

2. Primary Outcome: QOL-AD--PWD
Description: as for outcome 1
Time Frame: Week 12
Population: Overall number of participants analyzed corresponds to the number of participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 23
score on a scale | 35.23 (6.54) | 40.0 (5.36) | 36.68 (4.76) | 35.96 (8.04)

3. Secondary Outcome: Community Structure--PWD
Description: This is a brain imaging variable derived from fMRI images. Modularity (Q) ranges from 0 (no community structure) to 1 (perfectly modular network). One Q-value is generated for each person and group averages are shown.
Time Frame: Baseline
Population: Participants are missing at baseline imaging data due to an undisclosed contraindicated device, aborting scan, refusing scans, or excessive head motion.
Measure: Mean (Standard Deviation); unit: Q-Value
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 23 | 21
Q-Value | .74 (.05) | .72 (.05) | .73 (.05) | .74 (.04)

4. Secondary Outcome: Community Structure--PWD
Description: as for outcome 3
Time Frame: Week 12
Population: Numbers at baseline and week 12 differ due to withdrawals, poor data quality, and inability to complete scans.
Measure: Mean (Standard Deviation); unit: Q-Value
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 20 | 20 | 18 | 19
Q-Value | .74 (.04) | .73 (.05) | .75 (.04) | .75 (.03)

5. Secondary Outcome: Global Efficiency (eGlob)--PWD
Description: This is a brain imaging variable derived from fMRI images.Scale ranges from 0 (no long-range information processing) to 1 (maximal distributed processing). Decreased Eglob has been associated with aging, cognitive impairment, and depression.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 23 | 21
score on a scale | .19 (.02) | .18 (.03) | .19 (.03) | .19 (.03)

6. Secondary Outcome: Global Efficiency (eGlob)--PWD
Description: as for outcome 5
Time Frame: Week 12
Population: Number at baseline and follow-up differ due to withdrawals, poor data quality, participant refusal of procedure, inability to complete scan.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 20 | 20 | 18 | 19
score on a scale | .19 (.03) | .18 (.03) | .19 (.02) | .19 (.03)

7. Secondary Outcome: Local Efficiency (eLoc)--PWD
Description: Scale ranges from 0 (no local connectivity) to 1 (maximal local connectivity - all connections are local) and has been observed to change with cognitive impairment and depression.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 23 | 21
units on a scale | .59 (.03) | .57 (.04) | .59 (.03) | .58 (.04)

8. Secondary Outcome: Local Efficiency (eLoc)--PWD
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 20 | 20 | 18 | 19
units on a scale | .58 (.03) | .58 (.03) | .59 (.03) | .58 (.04)

9. Secondary Outcome: Path Length--PWD
Description: Refers to the number of edges that must be crossed to get from one node to another. Longer path length in people with AD has been associated with slower cognitive performance, beta amyloid deposition, and depression.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of Edges
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 23 | 21
Number of Edges | 5.29 (.58) | 5.69 (1.17) | 5.42 (.78) | 5.52 (.93)

10. Secondary Outcome: Path Length--PWD
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Number of Edges
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 20 | 20 | 18 | 19
Number of Edges | 5.30 (.93) | 5.61 (.80) | 5.36 (.54) | 5.54 (1.09)

11. Secondary Outcome: Fullerton Advanced Balance Scale (Overall Balance) PWD
Description: Fullerton Advanced Balance Scale (FAB) measures balance using 10 different performance-based tests (scored 0 worst - 4 best), including; standing with feet together and eyes closed, standing on a foam pad with eyes closed, walking while turning the head from side to side rhythmically, functional standing reach, turning around to the left and right, stepping up and over a 6-inch box, standing on one leg, and a test for postural reaction. The scale goes from 0-40 with 40 being the best outcome and a cutoff of <=25 for risk of falls.
Time Frame: Baseline
Population: One participant is missing baseline data due to a recording error during data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 24
score on a scale | 23.71 (8.22) | 27.88 (5.40) | 24.22 (6.32) | 26.79 (4.57)

12. Secondary Outcome: Fullerton Advanced Balance Scale (Overall Balance) PWD
Description: as for outcome 11
Time Frame: Week 12
Population: Number at baseline and week 12 differ due to withdrawals.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 23
score on a scale | 23.41 (8.57) | 29.95 (4.33) | 24.27 (6.26) | 26.78 (6.65)

13. Secondary Outcome: Falls Efficacy Scale - International (FES) PWD
Description: A 16-item scale to assess fear of falling where higher scores reflect a higher fear and risk of falling. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 27.54 (10.06) | 22.64 (4.86) | 26.07 (7.76) | 25.56 (8.65)

14. Secondary Outcome: Falls Efficacy Scale - International (FES) PWD
Description: as for outcome 13
Time Frame: Week 12
Population: Overall number of participants analyzed corresponds to the number of participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 23
score on a scale | 27.23 (10.38) | 21.73 (5.32) | 25.36 (5.27) | 28.09 (11.42)

15. Secondary Outcome: Neuropsychiatric Inventory Questionnaire (NPI-Q)
Description: The NPI is a reliable and valid structured interview designed to assess neuropsychiatric symptoms in person with dementia through a structured interview with the caregiver. The NPI includes questions about 12 domains of symptoms: delusions, hallucinations, agitation/aggression, depression, anxiety, elation/ euphoria, apathy, disinhibition, irritability, aberrant motor activity, sleep, and eating. For each, symptom severity is scored on a scale of 0-4, with 4 being the worst outcome and caregiver distress is scored on a scale from 0-5, with 5 being the worst outcome. The sum of all 12 domains is calculated. Severity scores are reported here with a range from 0-36 with a higher score reflecting greater symptom severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 6.83 (5.64) | 5.44 (4.44) | 6.85 (4.86) | 7.72 (6.13)

16. Secondary Outcome: NPI-Q
Description: as for outcome 15
Time Frame: Week 12
Population: Number at baseline and follow-up differ due to withdrawals and due to staff error during data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 21 | 22 | 22 | 23
score on a scale | 6.38 (5.48) | 5.22 (4.66) | 5.63 (5.71) | 8.39 (5.25)

17. Secondary Outcome: Geriatric Depression Scale
Description: The person with dementia will be asked to complete a screening tool for assessing depression. This test has 15 yes/no questions with a yes receiving 1 point for a depressive answer. A total score is calculated and will be on a scale from 0-15 with 0-4 indicating no depression, 5-10 suggestive of a mild depression, and 11+ suggestive of severe depression.
Time Frame: Baseline
Population: Results at baseline for this outcome represent all PWD who were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 2.17 (2.50) | 1.24 (1.05) | 2.37 (2.13) | 2.04 (2.28)

18. Secondary Outcome: Geriatric Depression Scale
Description: as for outcome 17
Time Frame: Week 12
Population: Overall number of participants analyzed corresponds to the number of participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 23
score on a scale | 2.27 (2.76) | 1.32 (1.36) | 1.68 (1.29) | 2.74 (3.54)

19. Secondary Outcome: Geriatric Anxiety Scale
Description: The Geriatric Anxiety Scale measures symptoms of anxiety in older adults. A single total score ranges from 0 (low anxiety) to 63 (high anxiety). Four cutoff scores have been provided by authors in the manuals: 0-7 (normal anxiety), 8-15 (mild-moderate anxiety), 16-25 (moderate-severe anxiety), and 26-63 (severe anxiety).
Time Frame: Baseline
Population: Results at baseline for this outcome represent all PWD who were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 3.71 (3.34) | 2.92 (2.06) | 4.04 (3.01) | 3.56 (3.31)

20. Secondary Outcome: Geriatric Anxiety Scale
Description: as for outcome 19
Time Frame: Week 12
Population: Overall number of participants analyzed corresponds to the number of participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 23
score on a scale | 3.64 (3.63) | 2.23 (1.57) | 3.64 (3.27) | 4.0 (4.65)

21. Secondary Outcome: Apathy Evaluation Scale--PWD
Description: The Apathy Evaluation Scale (AES) addresses characteristics of goal directed behavior that reflect apathy including behavioral, cognitive, and emotional indicators. A short form will be used that has been modified for use with people with dementia. This shortened version has 10 questions scored 1-4 with 4 being the positive outcome answer. The total score is calculated and on a scale of 10-40 with lower scores reflecting less apathy and thus a better outcome.
Time Frame: Baseline
Population: Results at baseline for this outcome represent all PWD who were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 21.83 (8.49) | 18.88 (6.23) | 19.74 (7.04) | 18.44 (7.53)

22. Secondary Outcome: Apathy Evaluation Scale--PWD
Description: as for outcome 21
Time Frame: Week 12
Population: One participant is missing follow-up data due to a recording error during data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale | 19.32 (9.89) | 19.0 (6.61) | 18.68 (6.24) | 22.87 (7.50)

23. Secondary Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: The eSPPB is a brief test of global mobility function with excellent test-retest and inter-examiner reliability; is sensitive to change; is safe, and is a robust predictor of future physical disability and death. To avoid ceiling effects, investigators will use an expanded version (eSPPB) that increases the difficulty of the standing balance task by asking participants to hold postures for 30 instead of 10 seconds, adds a one-leg stand, and adds a narrow walk. The resulting score is normally distributed, continuous, and shows greater sensitivity to change. Dementia patients have lower scores on the SPPB so a favorable outcome for this outcome measure would be a significantly higher score post treatment. The eSPPB is scored as a continuous measure with a minimum score of 0 and a maximum score of 3.0 where 3 is the best possible outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
score on a scale | 1.57 (.55) | 1.99 (.37) | 1.67 (.46) | 1.86 (.40)

24. Secondary Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: as for outcome 23
Time Frame: Week 12
Population: Number at baseline and follow-up differ due to withdrawals, staff error, participant unwilling to complete, and participant unable to complete test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 21 | 21
score on a scale | 1.62 (.57) | 1.98 (.39) | 1.66 (.44) | 1.88 (.50)

25. Secondary Outcome: Postural Sway--PWD
Description: Center of pressure displacement (area of the 95% confidence ellipse) using an AccuSway forceplate. Center of pressure displacement is one way to characterize postural sway. Increased postural sway is correlated with decreased balance in older adults and increased fall risk. Center of pressure displacement was measured using the area of the 95% confidence ellipse using an AccuSway forceplate. Higher numbers indicate greater levels of postural sway.
Time Frame: Baseline
Population: Number of participants analyzed at baseline differs due to technical error.
Measure: Mean (Standard Deviation); unit: centimeter squared
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 25 | 26 | 25
centimeter squared | 0.42 (0.37) | 0.37 (0.14) | 0.36 (0.21) | 0.49 (0.44)

26. Secondary Outcome: Postural Sway--PWD
Description: as for outcome 25
Time Frame: Week 12
Population: Numbers averaged at baseline and follow-up differ due to withdrawals, technical errors, safety concern, participant unwilling and participant unable to continue.
Measure: Mean (Standard Deviation); unit: centimeter squared
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 21 | 20 | 22 | 21
centimeter squared | 0.41 (0.22) | 0.38 (0.20) | 0.41 (0.26) | 0.52 (0.42)

27. Secondary Outcome: Gait Speed--PWD
Description: The time one takes to walk a specified distance on level surfaces over a short distance. 4m usual gait speed was measured as part of the eSPPB.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 24 | 25 | 27 | 25
seconds | 5.47 (1.55) | 4.61 (1.03) | 5.12 (1.39) | 4.66 (.85)

28. Secondary Outcome: Gait Speed--PWD
Description: as for outcome 27
Time Frame: Week 12
Population: Number at baseline and follow-up differ due to withdrawals, staff error, participant unwilling to complete and participant unable to complete.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 22 | 22 | 21 | 21
seconds | 5.51 (1.71) | 4.79 (.94) | 5.12 (1.06) | 4.77 (1.14)

29. Secondary Outcome: Gait Variability--PWD
Description: Stride time variability, which is calculated out of the mean and standard deviation of stride time, reflects the change in time elapsed between the first two contacts of two consecutive footfalls of the same foot over a number of gait cycles. Increased gait variability is associated with increased fall risk in older adults.
Time Frame: Baseline
Population: Subject numbers differ due to equipment failure, subjects withdrawing, subject inability to complete task, or lost to follow up.
Measure: Mean (Standard Deviation); unit: percentage of variability
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 21 | 22 | 23 | 23
percentage of variability | 3.41 (1.57) | 3.10 (1.68) | 3.44 (1.27) | 3.15 (1.07)

30. Secondary Outcome: Gait Variability--PWD
Description: as for outcome 29
Time Frame: Week 12
Population: Subject numbers differ due to equipment failure, technical error, subjects withdrawing, subject inability to complete task, or subject unwilling to complete task.
Measure: Mean (Standard Deviation); unit: percentage of variability
Arm/Group | Dance Group | Non-group Dance | Social Group | No Contact
Number analyzed (Participants) | 21 | 21 | 20 | 22
percentage of variability | 4.46 (2.88) | 2.71 (.75) | 3.45 (1.30) | 4.06 (4.15)

31. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: a measure of body fat based on height and weight that applies to adult men and women--PWD only
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Blood Pressure
Description: PWD only
Time Frame: Baseline, Week12
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Neuroticism-Extraversion-Openness Five-Factor Inventory (NEO-FFI)
Description: A measure of five domains of personality (neuroticism, extraversion, openness, agreeableness, and conscientiousness). A higher score on any scale indicates stronger presence of that trait. PWD only
Time Frame: Baseline
Reporting Status: Not Posted

34. Other Pre Specified Outcome: White Matter Lesion Burden
Description: The volume of white matter lesions is calculated using the Lesion Segmentation Toolbox. PWD only.
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Blood-based Stress Biomarkers (Covariate or Alternative Hypothesis)
Description: Social engagement may change biomarkers of stress relevant for interpreting outcomes. These stress biomarkers include cortisol and allostatic load, a composite measure of blood-based biomarkers associated with chronically elevated stress. PWD only
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Caregiver Quality of Life With the 36-item Short-Form Health (SF-36)--Covariate or Alternative Hypothesis
Description: The SF-36 consists of 36 questions assessing physical functioning, role functioning difficulties caused by physical problems, bodily pain, general health, vitality, social functioning, role functioning difficulties caused by emotional problems, and mental health. High scores are representative of a great health status and better outcomes, while low scores are representative of a poor health status.
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Caregiver Burden With Zarit Caregiver Burden Scale--Covariate or Alternative Hypothesis
Description: The Zarit Caregiver Burden Scale is administered in interview form to the caregiver. It consists of 22 questions scored 0-4 with 0=Never, 1=Rarely, 2=Sometimes, 3=Quite Frequently, 4=Nearly Always. The total score range is 0-88 with 88 being the worst possible outcome. 0-20 represents little or no burden on the caregiver, 21-40 represents mild to moderate burden, 41-60 represents moderate to severe burden, and 61-88 represents severe burden.
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through Week 12
Description: Persons with dementia (PWDs) and caregivers make up participant dyads for this study. The National Institutes for Health (NIH) requires adverse events to be collected on both participants within the dyad, so AEs for both are reported here.
Groups:
- Dance Group--PWD: The Dance Group will participate in 1-hour group improvisational dance lessons 2x/week for 12 weeks. Improvisational dance classes are grounded in 4 principles that shape the tone of the class and result in a sense of social belonging: non-judgment, non-competitiveness, curiosity, and playfulness. The following training strategies are used to maintain: active imagination, variability, and pacing.
  Dance Group: Active imagination refers to working with imagery and is crucial in improvisatory practice. Verbal auditory cues are used to create movement scenarios that cue or activate the motor imagination. Variability means the improvisational method does not aim to learn a specific movement pattern and habituate to it. Cues are delivered quickly, one after another. Within an average of two minutes, tasks requiring quicker decision-making are introduced. Pacing is the rate at which new movement prompts are presented. Quick changes in pace avoid defaulting to habitual responses, thereby facilitating new movement options. Participants cannot rely on copying another, memory, or anticipation to address the motor problem.
- Dance Group--Caregivers: Caregivers of the PWDs in the Dance Group--these participants are part of the dyad mentioned in the participant flow.
- Non-group Dance--PWD: The Non-group dance intervention is designed to capture the same dance movement and auditory stimuli as the group class without social interaction. Recordings of the dance instructor teaching a dance class will be played. This will ensure participants hear comparable music and receive comparable verbal auditory cues to prompt dance movements that students in the group class will hear, without interacting with other people. Improvisational dance is particularly suited for this means of delivery because the primary method of instruction is verbal auditory cueing. Participants will be asked to follow the same schedule as participants in the Dance Group arm and complete 2 one-hour dance sessions each week.
  Non-Group Dance: The caregiver will be asked to stay in the area while the subject is dancing. A video camera will be affixed in an upper corner of the room to record individual dance sessions. This recording will yield data that a trained student or staff member can view and code to document movement fidelity (e.g., that the person has responded to the dance prompts and for the purpose of comparing the amount of quality of movements that occur in individual vs. group dance settings). For the first two sessions, study staff would observe the full dance session from outside the room to be sure that instruction was clear and adherence was attained, and that no safety issues arise.
- Non-group Dance--Caregivers: Caregivers of the Non-group Dance PWDs--these participants are part of the dyad mentioned in the participant flow.
- Social Group--PWD: The social group will consist of improvisational party games to foster curiosity and playfulness, use imagery, and encourage non-judgment. Games that may be used include 'Balderdash', 'Wise and Otherwise', 'Charades', 'Pictionary', and 'Tell Me A Story' cards. These games will also use the same core strategies as the dance group. Games will be varied within an hour-long session to incorporate pacing and variability into the social group, akin to the dance group. The social group will occur 2x/week for 1 hour each time and be led by the same instructors who lead the Dance Group, to control for effects of personality of the group leader.
  Social Group: The social group will consist of improvisational party games to foster curiosity and playfulness, use imagery, and encourage non-judgment. Games that may be used include 'Balderdash', 'Wise and Otherwise', 'Charades', 'Pictionary', and 'Tell Me A Story' cards. These games will also use the same core strategies as the dance group. Games will be varied within an hour-long session to incorporate pacing and variability into the social group, akin to the dance group. The social group will occur 2x/week for 1 hour each time and be led by the same instructors who lead the Dance Group, to control for effects of personality of the group leader.
- Social Group--Caregivers: Caregivers of the Social Group PWDs--these participants are part of the dyad mentioned in the participant flow.
- No Contact--PWD: A No Contact condition captures the condition of no added social contact and no added dance movement. Participants randomized to the No Contact condition will be asked to continue their current disease management and lifestyle for 12 weeks
  No Contact: The condition of not receiving an intervention can have ethical implications and reduce retention rates. Therefore, these participants will be invited to join in a weekly community improvisational dance class after they complete the study, for as many sessions as they would like.
- No Contact--Caregivers: Caregivers of the No Contact PWDs--these participants are part of the dyad mentioned in the participant flow.
- Never Randomized-- PWD: PWD who dropped out before randomization
- Never Randomized--Caregiver: Caregivers of the PWDs who never randomized.
Arm/Group | Dance Group--PWD | Dance Group--Caregivers | Non-group Dance--PWD | Non-group Dance--Caregivers | Social Group--PWD | Social Group--Caregivers | No Contact--PWD | No Contact--Caregivers | Never Randomized-- PWD | Never Randomized--Caregiver
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/25 | 0/25 | 0/27 | 0/27 | 0/25 | 0/25 | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/24 | 4/24 | 0/25 | 2/25 | 2/27 | 4/27 | 4/25 | 2/25 | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 15/24 | 13/24 | 15/25 | 5/25 | 11/27 | 8/27 | 17/25 | 15/25 | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dance Group--PWD (N=24) | Dance Group--Caregivers (N=24) | Non-group Dance--PWD (N=25) | Non-group Dance--Caregivers (N=25) | Social Group--PWD (N=27) | Social Group--Caregivers (N=27) | No Contact--PWD (N=25) | No Contact--Caregivers (N=25) | Never Randomized-- PWD (N=3) | Never Randomized--Caregiver (N=3)
Heart attack (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrence (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elective full knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emergency room visit for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Admitted to hospital for suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
New diagnosis of non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in hip due to sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emergency room visit due to difficulty swallowing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fell walking across street and hit chest on sidewalk (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emergency room visit for chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidentally given dilaudid in hospital (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure due to COVID (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hit head falling backward getting out of bed (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Numbness and lack of coordination in arm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complications and infection from hernia surgery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (prior to randomization) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dance Group--PWD (N=24) | Dance Group--Caregivers (N=24) | Non-group Dance--PWD (N=25) | Non-group Dance--Caregivers (N=25) | Social Group--PWD (N=27) | Social Group--Caregivers (N=27) | No Contact--PWD (N=25) | No Contact--Caregivers (N=25) | Never Randomized-- PWD (N=3) | Never Randomized--Caregiver (N=3)
Sprained foot after fall (unrelated to study) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder pain from arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shingles (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall outside of study, no treatment needed (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 5 (6) | 0 (0) | 4 (5) | 4 (5) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Fall during data collection visit, no treatment needed (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stumbled at home (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulled muscle in lower back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain due to gastrointestinal issue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discontinued atorvastatin (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee and hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache, swollen jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip pain during intervention (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Side effects from donepezil (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Chest pain and dizziness (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slipped on wet pavement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exhaustion spell (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Broken ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Recurrent pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthroscopy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis flare (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration of thyroid nodule (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye surgery (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal lab results (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incidental finding on MRI-space occupying lesion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seen by surgeon for hernia surgery-no treatment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured patellar tendon (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labored breathing and chest pain when bending over (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth implants (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea and cough (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laser cytoscopy for bladder stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma removed from arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Admitted to rehabilitation center (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilateral recurrent inguinal hernia repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection in finger (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swimmer's ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injections for knee pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Removal of squamous cell carcinoma (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03333837/Prot_SAP_003.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03333837/ICF_002.pdf